CLINICAL TRIAL: NCT01378390
Title: Randomized, Single-blind, Placebo Controlled Multicenter Phase III Study to Assess the Efficacy and Safety of Expanded Autologous Adipose-derived Stem Cells (ASCs) (CX-401), for Treatment of Complex Perianal Fistulas in Perianal Crohn's Disease
Brief Title: Safety and Efficacy of Adipose-Derived Stem Cells to Treat Complex Perianal Fistulas Patients With Crohn's Disease
Acronym: FATT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: After the investigators and experts in the field imput it became apparent that the protocol was not reflective of clinical reality. No safety issues reported.
Sponsor: Tigenix S.A.U. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CX-401/FATT2; EudraCT: 2008-004286-25
Record Dates: First submitted 2011-06-21; First posted 2011-06-22 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Complex Perianal Fistula; Crohn Disease
Keywords: Complex perianal fistula; Crohn disease; Adipose-derived stem cells; Liposuction
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ASCs (Experimental): Intralesional dose of 20 million cells at baseline with a possible second administration of 40 million cells in case of incomplete fistula closure following week 12 assessment.
  Interventions: Drug: Expanded autologous adipose-derived adult stem cells (eASCs)
- Placebo (Sham Comparator): Instillation of saline solution into the fistulous tract, following identical tract preparation process as for the investigational treatment group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Expanded autologous adipose-derived adult stem cells (eASCs) — Administration will be preceded by localization and closure of the internal opening. Cell treatment injection will be performed following Major Ambulatory Surgery standards. Patients will receive an intralesional dose of 20 million cells at baseline. 50% of the cell suspension will be placed into the fistula walls of the internal opening, with the remaining 50% being injected across the wall tracts of the target fistula. Patients without healing (complete fistula closure) at week 12 will receive a second dose of 40 million cells, using the same treatment approach.
  Other Names: Cx401 (company code); Ontaril®
  Arms: ASCs
Drug: Placebo — Administration will be preceded by localization and closure of the internal opening following Major Ambulatory Surgery standards. Subjects will be receiving one treatment cycle with placebo consisting of intralesional instillation of 5 ml saline solution. Patients without healing (complete fistula closure) following week 12 assessment will continue to receive standard of care until the primary assessment of fistula closure at week 24. Patients with incomplete fistula closure at week 24 will be offered the possibility of participating in a separate open-label, single arm study using the ASCs derived from the liposuction procedure.
  Other Names: Normale saline solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine safety and efficacy of eASCs (expanded adult stem cells) for treatment of complex perianal fistulas in patients with Crohn's disease.

DETAILED DESCRIPTION:
Complex perianal fistulas are a source of great distress for suffers. In Crohn's disease, options are limited, and surgery is often associated with incontinence and recurrence.

The biological properties of stem cells derived from adult tissues make them candidates for the treatment of pathologies requiring tissue regeneration or in diseases where the healing process is altered.

A proof-of-concept study, a phase 1 study and a phase 2 study [Clinicaltrials.gov identifier: NCT00115466] have all suggested that this approach is promising, even in patients whose fistula is associated with Crohn's disease.

The present multicenter, placebo-controlled, phase 3 study aims to confirm the efficacy and safety shown in the previous phase 1 and phase 2 studies in the treatment of complex perianal fistulas in patients with Crohn's disease after 24 weeks from initial administration. Fistula closure is defined as absence of suppuration through the external orifice with complete re-epithelization of the external orifice and absence of collections >2cm directly related to the fistula tract treated, as measured by MRI.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patients with Crohn's disease diagnosed at least 12 months earlier in accordance with accepted clinical, endoscopic, anatomopathological and/or radiologic criteria
* Presence of complex perianal fistula with 3 or fewer fistulous tracts assessed by MRI
* Patients with persistent and active complex perianal fistula and non-active luminal Crohn's disease defined by a CDAI ≤ 200. (Complex perianal fistula is defined as a fistula that meets one or more of the following criteria: High fistulas [high inter-sphincteric, high trans-sphincteric, extra-sphincteric or supra-sphincteric], presence of 3 or fewer external openings [tracts] associated with a complex perianal fistula, or pain/fluctuation
* Good general state of health according to the findings of the clinical history and the physical examination
* Women of a childbearing age with negative serum or urine pregnancy test (sensitive to 25 IU hCG). Both men and women should use appropriate birth control methods defined by the investigator

Exclusion Criteria:

* Presence of severe proctitis (prominent friability, spontaneous bleeding, multiple erosions, deep ulcers) or dominant active luminal disease requiring immediate therapy, assessed by rectosigmoidoscopy
* Patients with a CDAI ≥201
* Patients with an abscess unless a complete toilet of the area with drainage of the collections and the absence of abscess and other collections is confirmed prior to treatment start
* The presence of setons unless removed prior to the study procedure
* Presence of >3 fistulous tracts and/or external openings
* Patients with rectal and/or anal stenosis evaluated by rectoscopy or EUA
* Patients who have received infliximab or any other anti-TNF agent in the 8 weeks before the cell treatment administration
* Patients who have received tacrolimus or cyclosporine in the 4 weeks before the cell treatment administration
* Patients with rectovaginal fistula, anal fistula(s), and/or non-perianal enterocutaneous fistula
* Patients with HIV, HBV, HCV or treponema infection, whether active or latent
* Patients with a history of abuse of alcohol or other addictive substances in the 6 months prior to inclusion
* Patients with malignant tumor, except for basal cell or cutaneous squamous cell carcinoma, or patients with a prior history of malignant tumors, unless the neoplastic disease has been in remission for the previous 5 years
* Patients with cardiopulmonary disease which, in the opinion of the investigator, is unstable or sufficiently serious to exclude the patient from the study.
* Patients with any type of medical or psychiatric disease which, in the opinion of the investigator, could be grounds for exclusion from the study
* Patients with congenital or acquired immunodeficiencies
* Patients with abnormal laboratory test findings that contraindicate their inclusion in the study
* Patients allergic to local anesthetics or gadolinium (MRI contrast)
* MRI is unfeasible, (e.g. due to the presence of pacemakers, hip replacements or severe claustrophobia)
* Liposuction with extraction of at least 100 cm3 of fat from the abdominal wall is technically unfeasible or the patient does not consent to the procedure
* Patients in need of surgery in the perianal region for reasons other than fistulas at the time of inclusion in the study, or a need for such surgery is foreseen in this region in the 26 weeks after treatment administration.
* Patients who have suffered major surgery or severe trauma in the prior 6 months
* Pregnant or breastfeeding women
* Patients who do not wish to or cannot comply with study procedures
* Patients currently receiving, or having received within 1 month prior to enrolment into this clinical trial, any investigational drug
* Patients unlikely to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects in whom the external openings of the treated perianal fistula have closed | 24 weeks

SECONDARY OUTCOMES:
Percentage of subjects in whom the external openings of the treated perianal fistula have closed | 12 weeks
Changes over time in the Perianal Disease Activity Index | 4, 10, 12, 16, 22 and 24 weeks
Changes over time in the Crohn's Disease Activity Index | 10 and 22 weeks
Changes over time in the MRI Score of Severity (MSS) | 12 and 24 weeks
Quality of life assessment using the SF-36 questionnaire | 12 and 24 weeks
Percentage of subjects for whom surgery is avoided | 24 weeks
Adverse events | 4, 10, 12, 16, 22 and 24 weeks
Clinically relevant variations in vital signs | 4, 10, 12, 16, 22 and 24 weeks
Clinically relevant variations in laboratory tests | 4, 10, 12, 16, 22 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Damián García-Olmo, MD, Principal Investigator — General Surgery Department, Hospital Universitario La Paz
Locations (12):
- University of Vienna, Vienna, Austria
- Academic Medical Center, Amsterdam, Netherlands
- Spain (10):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de Sagunto, Sagunto, Valencia
  - Hospital Reina Sofia, Córdoba
  - Complejo Hospitalario de León, Léon
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Complejo Hospitalario de Pontevedra, Pontevedra

REFERENCES:
- [Background] Garcia-Olmo D, Garcia-Arranz M, Garcia LG, Cuellar ES, Blanco IF, Prianes LA, Montes JA, Pinto FL, Marcos DH, Garcia-Sancho L. Autologous stem cell transplantation for treatment of rectovaginal fistula in perianal Crohn's disease: a new cell-based therapy. Int J Colorectal Dis. 2003 Sep;18(5):451-4. doi: 10.1007/s00384-003-0490-3. Epub 2003 May 20. PMID 12756590
- [Background] Garcia-Olmo D, Garcia-Arranz M, Herreros D, Pascual I, Peiro C, Rodriguez-Montes JA. A phase I clinical trial of the treatment of Crohn's fistula by adipose mesenchymal stem cell transplantation. Dis Colon Rectum. 2005 Jul;48(7):1416-23. doi: 10.1007/s10350-005-0052-6. PMID 15933795
- [Background] Garcia-Olmo D, Herreros D, Pascual M, Pascual I, De-La-Quintana P, Trebol J, Garcia-Arranz M. Treatment of enterocutaneous fistula in Crohn's Disease with adipose-derived stem cells: a comparison of protocols with and without cell expansion. Int J Colorectal Dis. 2009 Jan;24(1):27-30. doi: 10.1007/s00384-008-0559-0. Epub 2008 Aug 12. PMID 18696086
- [Background] Garcia-Olmo D, Garcia-Arranz M, Herreros D. Expanded adipose-derived stem cells for the treatment of complex perianal fistula including Crohn's disease. Expert Opin Biol Ther. 2008 Sep;8(9):1417-23. doi: 10.1517/14712598.8.9.1417. PMID 18694359